CLINICAL TRIAL: NCT03512951
Title: Subjective Evaluation of a Sound Externalization Method in Remote Microphone Systems for Binaural Hearing Aids With Respect to Auditory Distance Perception
Brief Title: Subjective Evaluation of a Sound Processing Method for Hearing Aids on Auditory Distance Perception
Acronym: EXTEND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Gilles Courtois (Unknown); Vincent Grimaldi (Unknown); Eleftheria Georganti (Unknown); Peter Derleth (Unknown); David Sooprayen (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ID 2018-00709
Record Dates: First submitted 2018-04-17; First posted 2018-05-01 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Hearing Disorders; Hearing Loss, Sensorineural
Keywords: Hearing aids; Remote microphone systems; Roger technology; Sound externalization; Auditory distance estimation
MeSH Terms: conditions — Hearing Disorders; Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal hearing (Experimental): A control group including ten normal-hearing participants. These participants are recruited because they can be considered as a reference when compared to hearing-impaired patients. They usually provide homogeneous results that are expected to be significantly different than those obtained with hearing-impaired patients. In this study, normal-hearing participants are expected to provide better and more consistent performance of auditory distance estimation.
  Interventions: Other: Digital signal processing algorithms
- 10 experienced hearing impaired (Experimental): A group of ten (expected sample size) severe-to-profound hearing-impaired patients who have a past and/or present experience of more than 6 months with remote microphone systems. These patients are expected to be aware of the drawbacks of the current remote microphone technology with respect to sound localization, auditory distance estimation, and audio-visual fusion.
  Interventions: Other: Digital signal processing algorithms
- 10 naive hearing impaired (Experimental): A group of ten severe-to-profound hearing-impaired patients with no past or current experience with remote microphone systems. They are referred to as naïve patients. These patients must have similar profiles to the patients in the experienced group as regards the degree of hearing loss, origin of hearing loss (congenital, pre- or post-lingual disability), age, gender, and hearing aid technology. They will be selected and recruited on the basis of the patients included in experienced group
  Interventions: Other: Digital signal processing algorithms

INTERVENTIONS:
Other: Digital signal processing algorithms — The intervention consists in applying five processing on some recorded speech signals. In particular, the processing performed by one specific algorithm is compared against the four other. The applied processing is supposed to restore sound externalization (expected audio-visual fusion).

SUMMARY:
Within the course of this study, a signal processing feature has been developed at Ecole Polytechnique Fédérale de Lausanne (EPFL), in collaboration with Sonova AG, in order to enhance the listening experience with remote microphone systems. In particular, the developed feature is supposed to improve the so-called audio-visual fusion, i.e. the fact to perceive the sound as coming from the physical location of the source. One of the main goals of the present study is to evaluate the extent to which this feature reaches that objective.

ELIGIBILITY:
Subjects fulfilling all of the following inclusion criteria are eligible for the study:

* Willing and able to give written informed consent as documented by signature,
* French-native adult speakers,
* (Preferably) younger than 60 y.o.

For all normal-hearing participants:

- Hearing thresholds lower or equal to 20 dB on both ears, as ensured by a pure-tone audiometry (125 Hz to 8 kHz) conducted at the beginning of the session.

For all hearing-impaired patients:

* Patients of Mr. Philippe Estoppey, private audiologist settled in Lausanne,
* User of bilateral BTE Phonak hearing aids, commercialized after July 2012, with fittings that did not change over the last three months,
* Presenting a severe-to-profound sensorineural hearing loss,
* Presenting a symmetrical hearing loss (no bilateral hearing threshold that differ by more than 20 dB at any audiometric frequency (125 Hz - 4 kHz)).

For HI patients experienced with remote microphone systems:

- Past or present users of FM and/or Roger devices for more than six months.

For other HI patients:

- No past or present experience with FM and/or Roger devices for more than one month.

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Collaborator of the laboratory (LTS2) or student attending the courses of audio and acoustics given by the laboratory staff (EE-348 Electroacoustics, EE-548 Audio Engineering),
* History of chronic or terminal illness, psychiatric disturbance, senile dementia, or cognitive impairment,
* History of strong tinnitus and/or hyperacusis,
* Strong visual impairment after correction with glasses or not,
* History of epilepsy or other reactions associated with the proximity to a screen,
* Motor disability that would disturb their presence at EPFL.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Auditory distance estimation | 6 months (study completion)
  This objective is assessed by using a single outcome, which is the perceived auditory distance, as reported by the patient on a graphical user interface. The auditory distance is measured using an arbitrary scale (between 1 and 5) as available with sliders on a graphical user interface (GUI).

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Ecole Polytechnique Fédérale de Lausanne, Lausanne, Canton of Vaud
  - Ecole Polytechnique Fédérale de Lausanne, Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Courtois G, Grimaldi V, Lissek H, Estoppey P, Georganti E. Perception of Auditory Distance in Normal-Hearing and Moderate-to-Profound Hearing-Impaired Listeners. Trends Hear. 2019 Jan-Dec;23:2331216519887615. doi: 10.1177/2331216519887615. PMID 31774032